CLINICAL TRIAL: NCT02415959
Title: A Phase II, Multicenter, Parallel-Group, Active-Controlled, Randomized, Double-blind, Dose-Ranging Study to Evaluate the Efficacy and Safety of Different Doses of Creon IR in Subjects With Pancreatic Exocrine Insufficiency Due to Cystic Fibrosis
Brief Title: Efficacy and Safety Study of Creon IR in Subjects With Pancreatic Exocrine Insufficiency Due to Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: AbbVie (Industry); LKF Laboratorium für Klinische Forschung GmbH (Unknown); Analytical Biochemical Laboratory (Unknown); Parexel (Industry); Datamap (Industry); Linical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: PANC2002; 2014-004519-35 (EudraCT Number)
Record Dates: First submitted 2015-03-19; First posted 2015-04-14 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Exocrine Pancreatic Insufficiency in Subjects With Cystic Fibrosis
Keywords: Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Creon IR low dose (Experimental): Creon IR 300 Ph. Eur. U lipase/g fat/day, proportionally administered five times daily (during 3 meals and 2 snacks) for 6 to 7 days (target total daily dose of 30,000 lipase units)
  Interventions: Drug: Creon IR
- Creon IR medium dose (Experimental): Creon IR 1,200 Ph. Eur. U lipase/g fat/day, proportionally administered five times daily (during 3 meals and 2 snacks) for 6 to 7 days (target total daily dose of 120,000 lipase units)
  Interventions: Drug: Creon IR
- Creon IR high dose (Experimental): Creon IR 2,400 Ph. Eur. U lipase/g fat/day, proportionally administered five times daily (during 3 meals and 2 snacks) for 6 to 7 days (target total daily dose of 240,000 lipase units)
  Interventions: Drug: Creon IR
- Creon IR maximum dose (Experimental): Creon IR 4,000 Ph. Eur. U lipase/g fat/day, proportionally administered five times daily (during 3 meals and 2 snacks) for 6 to 7 days (target total daily dose of 400,000 lipase units)
  Interventions: Drug: Creon IR
- Creon® (DR/GR) (Active Comparator): Creon® (DR/GR) 4,000 Ph. Eur. U lipase/g fat/day, proportionally administered five times daily (during 3 meals and 2 snacks) for 6 to 7 days (target total daily dose of 400,000 lipase units)
  Interventions: Drug: Creon® (DR/GR)

INTERVENTIONS:
Drug: Creon IR
  Arms: Creon IR high dose; Creon IR low dose; Creon IR maximum dose; Creon IR medium dose
Drug: Creon® (DR/GR)
  Arms: Creon® (DR/GR)

SUMMARY:
The objective of this study is to assess the efficacy and safety of different doses of Creon Immediate Release (IR) in comparison to Creon® 25,000 Delayed Release/Gastro-Resistant (DR/GR) in subjects with Pancreatic Exocrine Insufficiency (PEI) due to Cystis Fibrosis (CF).

DETAILED DESCRIPTION:
This study is a Phase II, randomized, parallel-group, active-controlled, double-blind, dose ranging, multicenter study with 4 different doses of Creon IR and one dose of the active control Creon® (DR/GR), administered in subjects of 12 years or older with PEI due to CF.

The study is divided into two periods: a screening period of 14 days and a double-blind treatment period of 6 to 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily signed and dated the Informed Consent Form (ICF). For subjects aged less than 18 years, the parents, or a legally acceptable representative, must sign consent and, as required by the Independent Ethics Committee (IEC), assent will be given by the subject.
2. Subject is 12 years old or older at the time of consent signature.
3. Subject has a diagnosis of CF previously confirmed by:

   * a sweat chloride test > or equal to 60 mmol/Ls and/or
   * two CF causing Cystic Fibrosis trans membrane conductance regulator (CFTR) mutations and
   * CF clinical features
4. Subject has a documented clinically confirmed diagnosis of pancreatic exocrine insufficiency.
5. Subject has human fecal elastase < 100 µg/g stool at screening
6. Subject has PEI that is currently clinically controlled (no clinically overt steatorrhea or diarrhea) under treatment with a commercially available Pancreatic enzyme Replacement Therapy (PERT), on an individually established dose regimen for more than 3 months, with a daily dose not exceeding 10,000 U lipase/kg/day.
7. Females of child-bearing potential and sexually active with men should agree to continue using a medically acceptable method of birth control throughout the study and for 7 days immediately after the last dose of study drug. Medically acceptable methods of birth control include bilateral tubal ligation or the use of either a contraceptive implant, a contraceptive injection (e.g., Depo Provera™), an intrauterine device, or an oral contraceptive taken continually within the past three months and which the subject agrees to continue using during the study or to adopt another birth control method, or a double-barrier method which consists of a combination of any two of the following: diaphragm, cervical cap, condom, or spermicide.

Exclusion Criteria:

1. Subject is < 18 years of age and has a Body Mass Index (BMI) Z-Score below -1.5 (minus 1.5)
2. Subject has a history of any of the following gastrointestinal disorders:

   * pancreatitis within 6 months prior to study entry;
   * fibrosing colonopathy;
   * distal ileal obstruction syndrome (DIOS) within 6 months prior to study entry;
   * celiac disease;
   * gastric bypass or partial/total gastrectomy;
   * Crohn's disease;
   * small bowel surgery (other than minor resection due to meconium ileus without resulting in malabsorption syndrome).
   * Any type of malignancy involving the digestive tract in the last 5 years.
3. Subjects with diabetes mellitus, for which the study specific dietary requirements may not be appropriate.
4. Subject has a history of other endocrine or respiratory (except mild asthma) medical illness non-related to CF, which might limit participation in or completion of the study.
5. Subject has a history of any clinically significant neurological, cardiac, renal, hepatic (including Hepatitis B or C), hematologic or psychiatric disease or disorder, or any other uncontrolled medical illness (except cystic fibrosis) which might limit participation in or completion of the study.
6. Subjects requiring concomitant treatment with any medication not allowed by the protocol or is expected to be needed.
7. Subjects requiring Naso-gastric, G-tubes or J-tubes.
8. Subject is currently participating in any other interventional clinical study or has taken any experimental drug within 30 days prior to Screening.
9. Subject is known to be HIV-positive.
10. Subject has a history of allergic reaction or significant sensitivity to pancreatin or inactive ingredients (excipients) of Creon® (DR/GR) or Creon IR

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suntje Sander-Struckmeier, PhD, Study Director — Abbott
Locations (17):
- Czechia (2):
  - Dětská nemocnice FN Brno, Centrum pro cystickou fibrozu, Brno
  - Klinika nemocí plicních a TBC, Brno
- Hungary (4):
  - Magyar Imre Kórház, Ajka
  - Kenézy Gyula Kórház, Debrecen
  - Kaposi Mór Oktató Kórház, Kaposvár
  - Tüdőgyógyintézet Törökbálint, Törökbálint
- Poland (5):
  - Centrum Medyczne Karpacz S.A., Karpacz
  - Wojewódzki Szpital Specjalistyczny Im M Kopernika W Łodzi, Lodz
  - Janusz Stankiewicz Sanatorium ""Cassia-Villa Medica, Rabka-Zdrój
  - Podkarpacki Ośrodek Pulmonologii i Alergologii, Rzeszów
  - ENEL-MED Szpital Centrum, Warsaw
- Spain (6):
  - Hospital Vall d ´Hebron, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Carlos Haya, Hospital Civil, Secretaria de Endocrinologia, Málaga
  - Hospital Universitario Virgen del Rocío, Hospital de la Mujer, Seville
  - Hospital La Fé Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Groups:
- Creon IR Low Dose: Creon IR 300 Ph. Eur. U lipase/g fat, proportionally administered five times daily (during 3 meals and 2 snacks) for 6 to 7 days (target total daily dose of 30,000 lipase units)
  Creon IR
- Creon IR Medium Dose: Creon IR 1,200 Ph. Eur. U lipase/g fat, proportionally administered five times daily (during 3 meals and 2 snacks) for 6 to 7 days (target total daily dose of 120,000 lipase units)
  Creon IR
- Creon IR High Dose: Creon IR 2,400 Ph. Eur. U lipase/g fat, proportionally administered five times daily (during 3 meals and 2 snacks) for 6 to 7 days (target total daily dose of 240,000 lipase units)
  Creon IR
- Creon IR Maximum Dose: Creon IR 4,000 Ph. Eur. U lipase/g fat, proportionally administered five times daily (during 3 meals and 2 snacks) for 6 to 7 days (target total daily dose of 400,000 lipase units)
  Creon IR
- Creon® (DR/GR): Creon® (DR/GR) 4,000 Ph. Eur. U lipase/g fat, proportionally administered five times daily (during 3 meals and 2 snacks) for 6 to 7 days (target total daily dose of 400,000 lipase units)
  Creon® (DR/GR)
Period: Overall Study
Arm/Group | Creon IR Low Dose | Creon IR Medium Dose | Creon IR High Dose | Creon IR Maximum Dose | Creon® (DR/GR)
Started | 14 | 14 | 14 | 14 | 14
Completed | 14 | 13 | 14 | 13 | 14
Not Completed | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Creon IR Low Dose | Creon IR Medium Dose | Creon IR High Dose | Creon IR Maximum Dose | Creon® (DR/GR) | Total
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 5 | 8 | 4 | 26
  Between 18 and 65 years | 10 | 9 | 9 | 6 | 10 | 44
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (7.6) | 22.9 (8.5) | 22.0 (7.3) | 19.7 (8.4) | 22.6 (7.1) | 22.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 7 | 5 | 6 | 33
  Male | 8 | 5 | 7 | 9 | 8 | 37
Region of Enrollment [Number; unit: participants]
  Hungary | 3 | 3 | 3 | 3 | 3 | 15
  Czech Republic | 1 | 1 | 1 | 1 | 1 | 5
  Poland | 6 | 6 | 6 | 6 | 6 | 30
  Spain | 4 | 4 | 4 | 4 | 4 | 20

OUTCOME MEASURES:

1. Primary Outcome: Coefficient of Fat Absorption (CFA)
Description: CFA is calculated from fat intake and fat excretion, according to the formula: CFA (%) = 100 [fat intake - fat excretion] / fat intake
Time Frame: End of the 6 to 7 days double-blind treatment period
Population: Full Analysis set. Four randomized subjects excluded because no post-baseline efficacy data (two non-completers and two subjects whose stools were mixed-up with each other at the analytical laboratory).
Measure: Mean (Standard Deviation); unit: percentage of fat intake
Arm/Group | Creon IR Low Dose | Creon IR Medium Dose | Creon IR High Dose | Creon IR Maximum Dose | Creon® (DR/GR)
Number analyzed (Participants) | 13 | 13 | 14 | 13 | 13
percentage of fat intake | 71.0 (12.4) | 70.9 (13.9) | 71.8 (15.2) | 75.9 (9.2) | 92.3 (3.7)

2. Secondary Outcome: Coefficient of Nitrogen Absorption (CNA)
Description: CNA is calculated from nitrogen intake and nitrogen excretion, according to the formula: CNA (%) = 100 [nitrogen intake - nitrogen excretion] / nitrogen intake)
Time Frame: End of the 6 to 7 days double-blind treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of nitrogen intake
Arm/Group | Creon IR Low Dose | Creon IR Medium Dose | Creon IR High Dose | Creon IR Maximum Dose | Creon® (DR/GR)
Number analyzed (Participants) | 13 | 13 | 14 | 13 | 13
percentage of nitrogen intake | 71.0 (10.0) | 73.2 (6.4) | 76.2 (8.1) | 79.9 (7.3) | 84.8 (4.3)

3. Secondary Outcome: Stool Fat Content
Description: Total amount of fat excreted during the stool collection period in grams.
Time Frame: End of the 6 to 7 days double-blind treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gram per 72 hours
Arm/Group | Creon IR Low Dose | Creon IR Medium Dose | Creon IR High Dose | Creon IR Maximum Dose | Creon® (DR/GR)
Number analyzed (Participants) | 13 | 13 | 14 | 13 | 13
gram per 72 hours | 87.5 (37.5) | 87.1 (41.0) | 84.1 (44.9) | 73.0 (28.2) | 23.5 (11.3)

4. Secondary Outcome: Stool Weight
Description: Total amount of stool weight during the collection period in grams
Time Frame: End of the 6 to 7 days double-blind treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gram per 72 hours
Arm/Group | Creon IR Low Dose | Creon IR Medium Dose | Creon IR High Dose | Creon IR Maximum Dose | Creon® (DR/GR)
Number analyzed (Participants) | 13 | 13 | 14 | 13 | 13
gram per 72 hours | 889.0 (294.2) | 905.3 (225.7) | 793.8 (279.8) | 755.7 (383.2) | 545.7 (256.3)

5. Other Pre Specified Outcome: Treatment Emergent Adverse Events
Description: Treatment emergent adverse events will be summarized per treatment group
Time Frame: From randomization to end of Double Blind period plus 1 day, i.e. up to 7/8 days
Measure: Number; unit: participants
Arm/Group | Creon IR Low Dose | Creon IR Medium Dose | Creon IR High Dose | Creon IR Maximum Dose | Creon® (DR/GR)
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14
participants | 10 | 9 | 7 | 9 | 7

ADVERSE EVENTS:
Arm/Group | Creon IR Low Dose | Creon IR Medium Dose | Creon IR High Dose | Creon IR Maximum Dose | Creon® (DR/GR)
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 1/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 10/14 | 9/14 | 7/14 | 9/14 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Creon IR Low Dose (N=14) | Creon IR Medium Dose (N=14) | Creon IR High Dose (N=14) | Creon IR Maximum Dose (N=14) | Creon® (DR/GR) (N=14)
infective pulmonary exacerbation due to CF (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Creon IR Low Dose (N=14) | Creon IR Medium Dose (N=14) | Creon IR High Dose (N=14) | Creon IR Maximum Dose (N=14) | Creon® (DR/GR) (N=14)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 8 (8) | 6 (6) | 4 (4) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2) | 6 (6) | 3 (3) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
faeces soft (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No